CLINICAL TRIAL: NCT05171686
Title: Association of Diuretics With Change in Extracellular Volume, Natriuretic Peptides, Symptoms, and Cardiovascular Outcomes in CKD
Brief Title: Diuretics and Volume Overload in Early CKD
Acronym: DOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEPH-001-21S; 1IK2CX002368-01A1 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-29 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: diuretic; chronic kidney disease; hypertension; extracellular volume; natriuretic peptides
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension | interventions — Hydrochlorothiazide; Chlorthalidone; Furosemide; Torsemide; Bumetanide

STUDY DESIGN:
Intervention Model Description: Open label single arm clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diuretic augmentation (Experimental): The participant's blood pressure medication regimen will be altered to initiate a thiazide-type or loop diuretic in those not already prescribed a diuretic, or to increase the dose if one is already prescribed.
  Interventions: Drug: Diuretic augmentation (hydrochlorothiazide, chlorthalidone, furosemide, torsemide, or bumetanide)

INTERVENTIONS:
Drug: Diuretic augmentation (hydrochlorothiazide, chlorthalidone, furosemide, torsemide, or bumetanide) — The participant's blood pressure medication regimen will then be altered to initiate a thiazide-type (hydrochlorothiazide or chlorthalidone) or loop diuretic (furosemide, bumetanide, or torsemide) in those not already prescribed a diuretic, or to increase the dose if one is already prescribed

SUMMARY:
Almost 15% of Americans have chronic kidney disease (CKD), with an even higher rate in Veterans due to common risk factors such as high blood pressure and diabetes. People with CKD have a high risk of cardiovascular (CV) diseases, such as heart attacks, heart failure, and strokes. Extra fluid in the body, called volume overload, may lead to CV disease in people with CKD. It is unknown if volume overload develops in the earliest stages of CKD, when treating it with common, inexpensive medicines called diuretics may improve long-term CV outcomes. This study will lay important groundwork to answer this question in Veterans with early CKD by comparing two ways to measure volume overload and studying the change in common symptoms like fatigue and short-term CV function after treatment with diuretic medicines.

DETAILED DESCRIPTION:
The investigators previously showed that brain natriuretic peptide (BNP) and N-terminal-pro-BNP (NT-pro-BNP), measures of ventricular stretch, are associated with death and cardiovascular (CV) outcomes in patients with chronic kidney disease (CKD) stages 1-3, and the investigators' preliminary pilot results suggest that these natriuretic peptides may correlate with objective measures of excess extracellular volume (ECV) and with symptoms common in CKD. The overarching objective is to determine if initiation of diuretic treatment or increase in dose is associated with changes in BNP and NT-pro-BNP, patient-reported symptom burden, and short-term hemodynamic parameters in patients with CKD stages 1-3 and elevated blood pressure, and whether these changes correlate with changes in ECV. The central hypothesis is that the change in ECV after starting or increasing diuretics in Veterans with stages 1-3 CKD is associated with changes in 1) natriuretic peptides, 2) patient-level factors, and 3) CV physiology.

The investigators will compare the changes in natriuretic peptides, symptoms, and CV parameters with the change in ECV after diuretic initiation or dose increase. The primary aim is to determine if initiation of diuretic treatment or increase in diuretic dose is associated with changes in natriuretic peptides. Secondary aims are to determine the effect of diuretic change on patient-reported symptom burden, and CV physiology.

This clinical trial will include 46 outpatients with CKD stages 1-3 and blood pressure >140/90 mmHg. At the first visit, the investigators will initiate or increase the dose of a thiazide or loop diuretic. Study measures other than echocardiogram will be repeated 4 weeks after the intervention to determine changes in these parameters. ECV will be measured by whole-body multifrequency bioimpedance spectroscopy (BIS), which is a validated, non-invasive, painless measure of ECV. Plasma BNP and NT-pro-BNP will be measured, and patient-reported fatigue, depression, and quality of life will be quantified using validated questionnaires. Hemodynamic parameters include blood pressure, pulse pressure, and total peripheral resistance index (TPRI) and cardiac index measured by Non-Invasive Hemodynamic Monitoring. A transthoracic echocardiogram will measure left ventricular mass index, valvular disease, and diastolic dysfunction.

Variables will be compared within participants between baseline and Visit 2 using paired Wilcoxon Signed Rank tests or paired Student's t tests, depending on variable distributions. Correlations between change in ECV/total body weight and all continuous outcome measures will be analyzed using Spearman or Pearson correlations, applying appropriate transformations. Linear regression analysis will control for clinically relevant variables. The relationship between ECV/total body weight and natriuretic peptides from both visits will be evaluated using a mixed effects model to account for the change in these measures between baseline and Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veterans age 18 years or older. There will be no upper age limit.
* The presence of CKD stages 1, 2, or 3, as defined below by Kidney Disease Improving Global Outcomes guidelines, for a period of at least 3 months.

  * Stage 1: eGFR 90 mL/min/1.73 m2 and spot urine albumin-to-creatinine ratio 30 mg/g.
  * Stage 2: eGFR 60-89 mL/min/1.73 m2 and spot urine albumin-to-creatinine ratio 30 mg/g.
  * Stage 3: eGFR 30-59 mL/min/1.73 m2.
* Measured blood pressure either >140 mmHg systolic or >90 mmHg diastolic at the two most recent clinic visits.
* Able to understand and sign informed consent after the nature of the study has been fully explained.

Exclusion Criteria:

* Unable to understand or provide informed consent.
* Unwilling or unable to participate in the protocol or comply with any of its components.
* CKD stages 4-5, defined as eGFR <30 mL/min/1.73 m2.
* Receiving chronic hemodialysis or peritoneal dialysis.
* Recipient of a kidney transplant.
* Serum potassium <3.5 mEq/L at baseline.
* Known left ventricular ejection fraction <40% on visual estimate based on chart review of available echocardiogram data.
* Known hepatic cirrhosis.
* Major limb amputation.
* Known pregnancy.
* Presence of a pacemaker or defibrillator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change in NT-pro-BNP | 4 weeks
  Change in NT-pro-BNP from baseline to 4 weeks after intervention

SECONDARY OUTCOMES:
Change in BNP | 4 weeks
  Change in BNP from baseline to 4 weeks after intervention
Change in FACIT-F score | 4 weeks
  Change in fatigue as measured by FACIT-F score from baseline to 4 weeks after intervention
Change in QIDS-SR16 | 4 weeks
  Change in depression as measured by the QIDS-SR16 from baseline to 4 weeks after intervention
Change in KDQOL | 4 weeks
  Change in quality of life as measured by the KDQOL from baseline to 4 weeks after intervention
Change in total peripheral resistance index | 4 weeks
  Change in total peripheral resistance index from baseline to 4 weeks after intervention
Change in systolic blood pressure | 4 weeks
  Change in systolic blood pressure from baseline to 4 weeks after intervention
Change in diastolic blood pressure | 4 weeks
  Change in diastolic blood pressure from baseline to 4 weeks after intervention
Change in mean arterial pressure | 4 weeks
  Change in mean arterial pressure from baseline to 4 weeks after intervention
Change in pulse pressure | 4 weeks
  Change in pulse pressure from baseline to 4 weeks after intervention
Change in cardiac index | 4 weeks
  Change in cardiac index from baseline to 4 weeks after intervention
Change in extracellular volume normalized/total body weight | 4 weeks
  Change in extracellular volume normalized to total body weight from baseline to 4 weeks after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lucile P Gregg, MD MS, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT05171686/ICF_001.pdf